CLINICAL TRIAL: NCT05754762
Title: Median Effective Dose of Remifentanil for the Prevention of Myoclonus Induced by Etomidate Injection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Zhuan Zhang, Director, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202230217
Record Dates: First submitted 2023-02-17; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Etomidate; Myoclonus
MeSH Terms: conditions — Myoclonus | interventions — Remifentanil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Age range of 18 to 40 years olds (Experimental): Based on previous literature and preliminary test results, the initial dose of pre-injection remifentanil is set at 1ug / kg. The dose of remifentanil is based on the patient's degree of myoclonus. If there is no myoclonus (negative response), the dose of remifentanil is reduced for the next patient until the patient develops myoclonus. If there is myoclonus (positive response), the dose of remifentanil will be increased in the next patient until the patient is free of myoclonus.
  Interventions: Drug: Remifentanil
- Age range of 41 to 55 years olds (Experimental): Based on previous literature and preliminary test results, the initial dose of pre-injection remifentanil is set at 1ug / kg. The dose of remifentanil is based on the patient's degree of myoclonus. If there is no myoclonus (negative response), the dose of remifentanil is reduced for the next patient until the patient develops myoclonus. If there is myoclonus (positive response), the dose of remifentanil will be increased in the next patient until the patient is free of myoclonus.
  Interventions: Drug: Remifentanil
- Age range of 56 to 70 years olds (Experimental): Based on previous literature and preliminary test results, the initial dose of pre-injection remifentanil is set at 1ug / kg. The dose of remifentanil is based on the patient's degree of myoclonus. If there is no myoclonus (negative response), the dose of remifentanil is reduced for the next patient until the patient develops myoclonus. If there is myoclonus (positive response), the dose of remifentanil will be increased in the next patient until the patient is free of myoclonus.
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — Advanced intravenous injection of remifentanil before the etomidate injection

SUMMARY:
Since its introduction in 1973, etomidate has been widely used in clinical anaesthesia, especially in haemodynamically unstable patients, as a new anaesthetic induction drug with the advantage of low circulatory and respiratory depression. When administered via intravenous injection, etomidate can cause adverse effects such as injection pain and myoclonus. The incidence of myoclonus is still reported to be as high as 50-80%. Myoclonus caused by etomidate may cause discomfort during induction of anaesthesia and reduce perioperative satisfaction, and may lead to syringe dislodgement, extravasation of the injected drug, swelling at the injection site, delayed induction of anaesthesia and, in severe cases, cardiovascular adverse events. Therefore, the myoclonus and limb retraction reactions caused by etomidate are a key concern for clinical anaesthesiologists and need to be addressed at a time when comfort anaesthesia is being promoted. The aim of this study was to reduce myoclonus produced by etomidate injection during induction of general anaesthesia in surgical patients and to investigate the half effective dose of remifentanil to reduce etomidate myoclonus.

ELIGIBILITY:
Inclusion Criteria:

1. Ages ranged from 18 to 80.
2. ASA # or # level.

Exclusion Criteria:

* Allergy or contraindication to remifentanil or rocuronium; required for Central venipuncture catheterization;
* Abnormal liver or kidney function;
* Heavy drinking and long-term use of sedatives, analgesics or anti-anxiety drugs;
* Hearing and language impairment;
* Peripheral vascular disease;
* Severe cardiovascular disease or neurological disorders;
* Failure of one-time peripheral venipuncture;
* Infection of hand or wrist skin.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
The presence of myoclonus | an average of 2 minutes
  Yes or No

SECONDARY OUTCOMES:
The levels of myoclonus | an average of 2 minutes